CLINICAL TRIAL: NCT00645372
Title: A Six Week, Multicenter, Double Blind, Double-Dummy, Parallel, Comparative Study To Compare The Efficacy, Safety And Tolerability Of Ziprasidone With Risperidone In The Treatment Of Chinese Subjects With Acute Exacerbation Of Schizophrenia
Brief Title: A Study to Compare the Efficacy and Safety of Ziprasidone and Risperidone for the Treatment of Schizophrenia in Chinese Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A1281115
Record Dates: First submitted 2008-03-24; First posted 2008-03-27 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone; ziprasidone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: Risperidone
- B (Experimental)
  Interventions: Drug: Ziprasidone

INTERVENTIONS:
Drug: Risperidone — Oral risperidone capsules 1 and 2 mg; doses were 1 mg once daily on Days 1-2, 2 mg once daily on Days 3-4, 3 mg once daily on Days 5-7, and 1, 2, or 3 mg twice daily during Weeks 2-6
  Arms: A
Drug: Ziprasidone — Oral ziprasidone capsules 40, 60, and 80 mg; doses were 40 mg twice daily on Days 1-2, 60 mg twice daily on Days 3-7, and 40, 60, or 80 mg twice daily during Weeks 2-6
  Arms: B

SUMMARY:
The purpose of this study is to compare the efficacy and safety of ziprasidone and risperidone for the treatment of schizophrenia in Chinese patients

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with schizophrenia
* Miminum PANSS score of 60 when randomized

Exclusion Criteria:

* Planned, regular use of antipsyhotics within 1 week of randomization
* Previous treatment with risperidone that resulted in intolerance or lack of response to risperidone

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2004-07; Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Positive and Negative Syndrome Scale (PANSS) total score | Week 6

SECONDARY OUTCOMES:
Adverse events, laboratory test changes, movement disorder scale scores | Weeks 1, 2, 4, and 6
Change from baseline in PANSS negative subscale score | Weeks 1, 2, 4, and 6
Change from baseline in PANSS general psychopathology subscale score | Weeks 1, 2, 4, and 6
PANSS responder rate | Weeks 1, 2, 4 and 6
Clinical Global Impression-Severity (CGI-S) score | Baseline and Weeks 1, 2, 4, and 6
Change from baseline in Brief Psychiatric Rating Scale derived (BPRSd) score | Weeks 1, 2, 4, and 6
Change from baseline in PANSS positive subscale score | Weeks 1, 2, 4, and 6
Clinical Global Impression-Improement (CGI-I) score | Weeks 1, 2, 4, and 6

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- China (4):
  - Pfizer Investigational Site, Beijing
  - Pfizer Investigational Site, Guangzhou
  - Pfizer Investigational Site, Nanjing
  - Pfizer Investigational Site, Shanghai

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1281115&StudyName=A%20study%20to%20compare%20the%20efficacy%20and%20safety%20of%20ziprasidone%20and%20risperidone%20for%20the%20treatment%20of%20schizophrenia%20in%20Chinese%20patients